CLINICAL TRIAL: NCT05251363
Title: BIOTRONIK Conduction System Pacing With the Solia Lead
Acronym: BIO-CONDUCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biotronik, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: G210349
Record Dates: First submitted 2022-02-07; First posted 2022-02-22 (Actual); Results first posted 2025-03-18 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-02

CONDITIONS: Bradycardia; Atrioventricular Block; Left Bundle-Branch Block; Cardiomyopathies
MeSH Terms: conditions — Bradycardia; Atrioventricular Block; Bundle-Branch Block; Cardiomyopathies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Solia S LBB lead (Other)
  Interventions: Device: Solia S lead

INTERVENTIONS:
Device: Solia S lead — The Solia S pacing lead will be implanted in the LBB area for patients who meet all inclusion/exclusion criteria and give written informed consent.

SUMMARY:
The purpose of the BIO-CONDUCT study is to demonstrate the safety and effectiveness of the BIOTRONIK Solia S pacing lead when implanted in the left bundle branch (LBB) area. Safety will be assessed by evaluating serious adverse device effects that occur through 3 months post-implant. Efficacy will be assessed by evaluating implant success rate.

ELIGIBILITY:
Inclusion Criteria:

* Patient is a candidate for implantation of a BIOTRONIK pacemaker system, per standard guidelines. Single chamber, dual chamber, and Cardiac Resynchronization Therapy with a Pacemaker (CRT-P) systems are allowed.
* Patient has an implant planned to utilize left bundle branch area pacing within 30 days of consent
* Patient is able to understand the nature of the study and provide written informed consent
* Patient is available for follow-up visits on a regular basis for the expected duration of follow-up
* Patient accepts Home Monitoring® concept
* Patient age is greater than or equal to 18 years at time of consent

Exclusion Criteria:

* Patient meets a standard contraindication for pacemaker system implant
* Patient is currently implanted with a pacemaker or Implantable Cardioverter-Defibrillator (ICD) device
* Patient has had a previous unsuccessful attempt to place a lead in the LBB area
* Patient has planned cardiac surgical procedures or interventional measures within 3 months after implant
* Patient is expected to receive a heart transplant within 12 months
* Patient life expectancy less than 12 months
* Patient has the presence of another life-threatening, underlying illness separate from their cardiac disorder
* Patient reports pregnancy at the time of enrollment
* Patient is enrolled in any other investigational cardiac clinical study during the course of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 194 (Actual)
Dates: Start 2022-12-12 (Actual); Primary Completion 2024-01-09 (Actual); Study Completion 2024-10-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (14):
- United States (14):
  - Banner - University Medical Center Phoenix, Phoenix, Arizona
  - Cardiology Associates Medical Group, Ventura, California
  - Washington Hospital Center, Washington D.C., District of Columbia
  - Sarasota Memorial Health Care System, Sarasota, Florida
  - Tampa General Hospital, Tampa, Florida
  - Rush University Medical Center, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Cardiology Associates, Tupelo, Mississippi
  - NYU Langone Health, New York, New York
  - Weill Cornell Medicine, New York, New York
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Cardiology Consultants of Philadelphia, Philadelphia, Pennsylvania
  - Geisinger, Wilkes-Barre, Pennsylvania
  - Medical University of South Carolina (MUSC), Charleston, South Carolina

IPD SHARING:
Plan to Share IPD: Yes
De-identified participant level data collected within the study will be shared for approved requests.
Supporting Information: Study Protocol, SAP
Time Frame: The data will be available beginning no later than 12 months and ending 3 years after study.
Access Criteria: Proposals should be directed to BIOTRONIK Clinical Studies (BIOTRONIK Inc., Attn: Clinical Studies, 6024 Jean Road, Lake Oswego, OR; 1-800-547-0394). BIOTRONIK, in consultation with the National Principal Investigator, will review and critique requests for scientific merit, fiscal feasibility, and logistical feasibility. If approved, the data requestors will need to sign a data use/access agreement prior to obtaining the data. BIOTRONIK reserves the right to delete any confidential information or other proprietary information (including trade secrets and patent protected materials) from the shared information.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first study subject was consented on December 12, 2022. Study enrollment was completed on September 22, 2023, with a total of 194 subjects consented at 14 sites.
Pre-assignment Details: Of the 194 enrolled participants, 186 met inclusion criteria and underwent an implant procedure attempt.
Groups:
- Solia S LBB Lead: Solia S lead: The Solia S pacing lead will be implanted in the LBBA for patients who meet all inclusion/exclusion criteria and give written informed consent.
Period: Implant
Arm/Group | Solia S LBB Lead
Started | 186 (Total subjects with an implant attempt)
Completed | 178 (Subjects with a successful LBBA implant (per protocol defined criteria))
Not Completed | 8
Not completed — Subject did not meet LBBA implant criteria | 8
Period: Overall Study After Implant Period
Arm/Group | Solia S LBB Lead
Started | 178
Protocol Follow-Up: 3-Month | 167
Protocol Follow-Up: 6-Month | 163
Protocol Follow-Up (Final): 12-Month | 155
Completed | 155
Not Completed | 23
Not completed — Death | 9
Not completed — Solia S lead in LBBA Position Extracted | 4
Not completed — Withdrawal by Subject | 4
Not completed — Lost to Follow-up | 2
Not completed — Physician Decision | 1
Not completed — Subject Moved from Investigational Center | 3

BASELINE CHARACTERISTICS:
Groups:
- Subjects With a Successful Solia S Implant in the LBBA: This includes subjects that were consented and had a successful Solia S LBBA lead implant according to the study implant success criteria.
Arm/Group | Subjects With a Successful Solia S Implant in the LBBA
Number analyzed (Participants) | 178
Age, Continuous [Mean (Standard Deviation); unit: Years] | 76.2 (9.12)
Sex: Female, Male [Count of Participants; unit: Participants] — The measure used is the sex at birth
  Participants
    Female | 65
    Male | 113
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8
  Not Hispanic or Latino | 156
  Unknown or Not Reported | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 15
  White | 142
  More than one race | 1
  Unknown or Not Reported | 17
Height [Mean (Standard Deviation); unit: Inches] — Population: Height data was provided by only 175 subjects.
  Inches
    number analyzed (Participants) | 175
    (all) | 67.4 (4.23)
Weight [Mean (Standard Deviation); unit: Pounds] — Population: Weight data was provided by only 176 subjects.
  Pounds
    number analyzed (Participants) | 176
    (all) | 186.3 (41.66)
BMI [Mean (Standard Deviation); unit: kg/m²] — Population: Height data (a component of BMI calculation), was provided by only 175 subjects.
  kg/m²
    number analyzed (Participants) | 175
    (all) | 28.8 (5.43)
Medical History [Count of Participants; unit: Participants]
  Heart Failure | 44
  Cardiomyopathy | 13
  Coronary Artery Disease | 61
  Prior Myocardial Infarction | 22
  Atrial Fibrillation | 81
  Diabetes Mellitus | 41
  Hypertension | 152
  Sleep Apnea | 47
  Chronic Obstructive Pulmonary Disease | 23
  Cerebrovascular Disease (e.g., TIA / Stroke) | 33
  Chronic Kidney Disease (CKD) | 44
  Valvular Heart Disease | 46
  Peripheral Artery Disease | 16
Cardiac Medication at Implant [Count of Participants; unit: Participants]
  ACE Inhibitors | 36
  Angiotensin Receptor Blocker | 51
  Angiotensin Receptor-Neprilisyn Inhibitor | 2
  Class I Antiarrhythmic/Sodium-channel Blocker | 9
  Class II Antiarrhythmic/Beta Blocker | 55
  Class III Antiarrhythmic/Potassium-channel Blocker | 15
  Class IV Antiarrhythmic/Calcium Channel Blocker | 40
  Digitalis | 2
  Anticoagulant | 68
  Antiplatelet | 57
  Aldosterone Antagonist | 6
  Diuretics Other Than Aldosterone Antagonist | 60
Implant Indication [Count of Participants; unit: Participants]
  Sinus Node Disease/Sick Sinus Syndrome | 87
  Atrioventricular (AV) Block | 70
  Planned or Prior AV Node Ablation | 9
  Primary Heart Failure Indication | 1
  Other | 11

OUTCOME MEASURES:

1. Primary Outcome: Serious Adverse Device Effect (SADE)-Free Rate at 3 Months
Description: The overall rate of serious Solia S Left Bundle Branch (LBB) lead related adverse device effects and serious implant procedure events related to the Solia S LBB lead that occur through 3 months post-implant. The definition of adverse device effect is an untoward medical occurrence (e.g. disease, injury) related to the use of a study device. Pacemaker lead-related examples include events such as lead dislodgements or lead malfunction. The Solia S LBB lead complication-free rate is calculated as the number of subjects without one or more adverse device effect complications divided by the total number of study subjects successfully enrolled and subjects undergoing an unsuccessful implant attempt who have a qualifying primary safety endpoint event. Classification of adverse device related events from the pool of potential events is determined by a clinical events committee (CEC). The complication-free rate is expressed in percent.
Time Frame: 3 months post implant
Population: BIO-CONDUCT (NCT05251363) intent-to-treat subjects (having a successful or attempted Solia S implant in the LBBA) or subjects who had a qualifying primary safety endpoint event (such as a disease or injury related to the use of Solia S in the LBBA) prior to their exit from the study, were pooled with subjects in the BIO|MASTER.Selectra 3D study (NCT04323670) who satisfied the BIO-CONDUCT inclusion/exclusion criteria and experienced the primary endpoint or had at least 76 days of follow-up.
Measure: Number (95% Confidence Interval); unit: Percentage of participants without SADE
Groups:
- Intent-to-treat (ITT) - Primary Endpoint 1: This group includes all enrolled subjects (subjects with successfully implanted Solia S in the LBBA) and subjects with an unsuccessful implant attempt of the Solia S in the LBBA who had a qualifying primary safety endpoint event prior to their exit from the study.
Arm/Group | Intent-to-treat (ITT) - Primary Endpoint 1
Number analyzed (Participants) | 178
Percentage of participants without SADE | 98 [95.4 to 99.3]
Statistical Analysis 1: Comparison: Intent-to-treat (ITT) - Primary Endpoint 1; Ho: SADE-free rate ≤ 87.5% Ha: SADE-free rate > 87.5% Used an exact binomial test comparing the observed proportion (overall SADE-free rate through 3 months) to the performance goal of 87.5%. The lower, two-sided 95% confidence bound for the overall SADE-free rate must be greater than 87.5% to reject the null hypothesis (Ho), which would demonstrate evidence that the SADE-free rate is significantly higher than 87.5%; Test type: Superiority; p < 0.0001, Exact binomial test

2. Primary Outcome: Implant Success Rate of the Solia S Lead in LBB Area
Description: The percentage of subjects with Solia S placed successfully in the LBBA divided by the total number of consented study subjects in whom an implant of Solia S in the LBBA was attempted.
Time Frame: at implant procedure
Population: The population is defined as all enrolled subjects (subjects with successfully implanted Solia S in the LBBA) and subjects with an unsuccessful implant attempt of the Solia S in the LBBA. Determination of implant success is defined by the implanting physician at time of implant and includes assessments of the correct lead placement in the LBBA area during lead fixation. Final lead position is confirmed again after fixation.
Measure: Number (95% Confidence Interval); unit: % of participants with implant success
Groups:
- Intent-to-Treat (ITT) - Primary Endpoint 2 (Efficacy): This group is defined as all enrolled subjects (subjects with successfully implanted Solia S in the LBBA) and subjects with an unsuccessful implant attempt of the Solia S in the LBBA.
Arm/Group | Intent-to-Treat (ITT) - Primary Endpoint 2 (Efficacy)
Number analyzed (Participants) | 186
% of participants with implant success | 95.7 [91.7 to 98.1]
Statistical Analysis 1: Comparison: Intent-to-Treat (ITT) - Primary Endpoint 2 (Efficacy); H0: Implant Success Rate ≤ 80% Ha: Implant Success Rate > 80% Used an exact binomial test comparing the observed proportion (implant success rate) to the performance goal of 80%. The lower, two-sided 95% confidence bound for the overall implant success rate must be greater than 80% to reject the null hypothesis (Ho), which would demonstrate evidence that the rate of successful Solia S LBBA implants is significantly higher than 80.0%; Test type: Superiority; p < 0.0001, Exact binomial test

3. Secondary Outcome: Quality of Life (QOL) From Baseline Through 12 Months Post-Implant
Description: The change in the physical function Short Form-36 (SF-36, 36-Item Short Form Health Survey) QOL subscale was calculated as the mean change from baseline to 12-month follow-up for all subjects that completed both the baseline QOL and 12-month QOL questionnaire. The physical function subscale of Short Form-36 is comprised of ten questions out of the total of 36 questions. The responses to the ten questions relating to physical function were averaged at baseline and at 12 months. The difference in the averages (12 months minus baseline) is reported as the outcome for secondary endpoint 1. Note that each question and each component is scored such that a higher score defines a more favorable health state. Each is scored on a 0 to 100 range so that the lowest and highest possible scores are 0 and 100, respectively.
Time Frame: 12 months post implant
Population: Population is defined as all enrolled subjects (subjects with successfully implanted Solia S in the LBBA) with evaluable, paired baseline and 12-mo measurements. Excludes subjects if baseline or 12-month QOL score cannot be calculated (due to missing or incomplete QOL data).
Measure: Mean (95% Confidence Interval); unit: Score on a Scale
Groups:
- Intent-to-Treat (ITT) - Secondary Endpoint 1 (QOL): This group is defined as all enrolled subjects (subjects with successfully implanted Solia S in the LBBA).
Arm/Group | Intent-to-Treat (ITT) - Secondary Endpoint 1 (QOL)
Number analyzed (Participants) | 139
Score on a Scale | 11.4 [7.4 to 15.4]
Statistical Analysis 1: Comparison: Intent-to-Treat (ITT) - Secondary Endpoint 1 (QOL); H0: Improvement in QOL Physical Function Scale ≤ 2.8 Ha: Improvement in QOL Physical Function Scale > 2.8 Exact one-sample t-test comparing mean improvement in QOL from baseline to 12-mo post-implant to a goal of +2.8. The lower, two-sided 95% confidence bound for the improvement in QOL must be > +2.8 to reject H0; Test type: Superiority; p < 0.001, t-test, 2 sided

4. Secondary Outcome: Serious Adverse Device Effect (SADE)-Free Rate at 6 Months
Description: The overall rate of serious Solia S LBBA lead related adverse device effects and serious implant procedure events related to the Solia S LBBA lead that occur through 6 months post-implant. The Solia S LBBA lead complication-free rate per subject, which was calculated as the number of subjects without one or more complications divided by the total number of study subjects successfully enrolled and subjects undergoing an unsuccessful implant attempt who have a qualifying safety endpoint event. The complication-free rate is expressed in percentage of participants without SADE.
Time Frame: 6 months post implant
Population: Descriptive analysis of BIO-CONDUCT (NCT05251363) intent-to-treat subjects (have a successfully implanted Solia S in the LBBA or had an unsuccessful implant attempt of Solia S in the LBBA) or subjects who had a qualifying primary safety endpoint event prior to their exit from the study were pooled with subjects in the BIO|MASTER.Selectra 3D study (NCT04323670) who satisfied the BIO-CONDUCT inclusion/exclusion criteria and experienced the primary endpoint or had at least 152 days of follow-up.
Measure: Mean (95% Confidence Interval); unit: Percentage of participants without SADE
Groups:
- Intent-to-Treat (ITT) - Secondary Endpoint 2 (SADE-Free Rate at 6-Mo): This group includes all enrolled subjects (subjects with successfully implanted Solia S in the LBBA) and subjects with an unsuccessful implant attempt of the Solia S in the LBBA who had a qualifying primary safety endpoint event prior to their exit from the study.
Arm/Group | Intent-to-Treat (ITT) - Secondary Endpoint 2 (SADE-Free Rate at 6-Mo)
Number analyzed (Participants) | 168
Percentage of participants without SADE | 96.7 [93.7 to 98.6]

5. Secondary Outcome: Serious Adverse Device Effect (SADE)-Free Rate at 12 Months
Description: The overall rate of serious Solia S LBBA lead related adverse device effects and serious implant procedure events related to the Solia S LBBA lead that occur through 12 months post-implant. The Solia S LBBA lead complication-free rate per subject, which was calculated as the number of subjects without one or more complications divided by the total number of study subjects successfully enrolled and subjects undergoing an unsuccessful implant attempt who have a qualifying safety endpoint event. The complication-free rate is expressed in percent.
Time Frame: 12 months post implant
Population: BIO-CONDUCT (NCT05251363) intent-to-treat subjects (have a successfully implanted Solia S in the LBBA or had an unsuccessful implant attempt of the Solia S in the LBBA) or subjects who had a qualifying primary safety endpoint event prior to their exit from the study were pooled with subjects in the BIO|MASTER.Selectra 3D study (NCT04323670) who satisfied the BIO-CONDUCT inclusion/exclusion criteria and experienced the primary endpoint or had at least 335 days of follow-up.
Measure: Mean (95% Confidence Interval); unit: Percentage of participants without SADE
Groups:
- Intent-to-Treat (ITT) - Secondary Endpoint 2 (SADE-Free Rate at 12-Mo): This group includes all enrolled subjects (subjects with successfully implanted Solia S in the LBBA) and subjects with an unsuccessful implant attempt of the Solia S in the LBBA who had a qualifying primary safety endpoint event prior to their exit from the study.
Arm/Group | Intent-to-Treat (ITT) - Secondary Endpoint 2 (SADE-Free Rate at 12-Mo)
Number analyzed (Participants) | 161
Percentage of participants without SADE | 96.1 [92.6 to 98.2]

6. Secondary Outcome: Pacing Threshold Measurements for Solia S Lead at 3 Months
Description: Pacing threshold measurements for Solia S leads implanted in the LBBA at the 3 month follow-up visit.
Time Frame: 3 months post implant
Population: Includes Intent-to-Treat (ITT) subjects with valid threshold measurements at their 3-mo follow-up. Some leads may not have a value at a visit due to valid reasons, such as remote threshold information (capture control or automatic threshold measurement) is not available or thresholds not being performed at 0.4 ms, or due to source documentation being unavailable.
Measure: Mean (Standard Deviation); unit: Volts @ 0.4ms
Groups:
- Intent-to-Treat (ITT) - Secondary Endpoint 3 (Pacing Threshold at 3-Mo): All enrolled subjects (subjects with successfully implanted Solia S in the LBBA)
Arm/Group | Intent-to-Treat (ITT) - Secondary Endpoint 3 (Pacing Threshold at 3-Mo)
Number analyzed (Participants) | 156
Volts @ 0.4ms | 0.94 (0.26)

7. Secondary Outcome: Sensing Measurements for Solia S Lead at 3 Months
Description: R-wave sensing amplitude measurements for Solia S leads implanted in the LBBA at the 3 month follow-up visit.
Time Frame: 3 months post implant
Population: Includes Intent-to-Treat (ITT) subjects with valid R-wave sensed amplitude measurements at their 3-mo follow-up. Some leads may not have a value at a visit due to valid reasons, such as atrial fibrillation or complete heart block, or due to source documentation being unavailable.
Measure: Mean (Standard Deviation); unit: mV
Groups:
- Intent-to-Treat (ITT) - Secondary Endpoint 4 (R-wave Sensed Amplitude at 3-Mo): All enrolled subjects (subjects with successfully implanted Solia S in the LBBA)
Arm/Group | Intent-to-Treat (ITT) - Secondary Endpoint 4 (R-wave Sensed Amplitude at 3-Mo)
Number analyzed (Participants) | 162
mV | 12.37 (4.16)

8. Secondary Outcome: Pacing Impedance for Solia S Lead at 3 Months
Description: Pacing impedance measurements for Solia S leads implanted in the LBBA at the 3 month follow-up visit.
Time Frame: 3 months post implant
Population: Includes Intent-to-Treat (ITT) subjects with valid pacing impedance measurements at their 3-mo follow-up. Some leads may not have a value at a visit due to valid reasons such as remote due to source documentation being unavailable
Measure: Mean (Standard Deviation); unit: Impedance (Ω)
Groups:
- Intent-to-Treat (ITT) - Secondary Endpoint 5 (Pacing Impedance at 3-Mo): All enrolled subjects (subjects with successfully implanted Solia S in the LBBA)
Arm/Group | Intent-to-Treat (ITT) - Secondary Endpoint 5 (Pacing Impedance at 3-Mo)
Number analyzed (Participants) | 166
Impedance (Ω) | 540.4 (96.4)

9. Secondary Outcome: Pacing Threshold Measurements for Solia S Lead at 6 Months
Description: Pacing threshold measurements for Solia S leads implanted in the LBBA at the 6 month follow-up visit.
Time Frame: 6 months post implant
Population: Includes Intent-to-Treat (ITT) subjects with valid threshold measurements at their 6-mo follow-up. Some leads may not have a value at a visit due to valid reasons, such as remote threshold information (capture control or automatic threshold measurement) is not available or thresholds not being performed at 0.4 ms, or due to source documentation being unavailable.
Measure: Mean (Standard Deviation); unit: Volts @ 0.4ms
Groups:
- Intent-to-Treat (ITT) - Secondary Endpoint 3 (Pacing Threshold at 6-Mo): All enrolled subjects (subjects with successfully implanted Solia S in the LBBA)
Arm/Group | Intent-to-Treat (ITT) - Secondary Endpoint 3 (Pacing Threshold at 6-Mo)
Number analyzed (Participants) | 146
Volts @ 0.4ms | 0.97 (0.27)

10. Secondary Outcome: Sensing Measurements for Solia S Lead at 6 Months
Description: R-wave sensing amplitude measurements for Solia S leads implanted in the LBBA at the 6 month follow-up visit.
Time Frame: 6 months post implant
Population: Includes Intent-to-Treat (ITT) subjects with valid R-wave sensed amplitude measurements at their 6-mo follow-up. Some leads may not have a value at a visit due to valid reasons, such as atrial fibrillation or complete heart block, or due to source documentation being unavailable.
Measure: Mean (Standard Deviation); unit: mV
Groups:
- Intent-to-Treat (ITT) - Secondary Endpoint 4 (R-wave Sensed Amplitude at 6-Mo): All enrolled subjects (subjects with successfully implanted Solia S in the LBBA)
Arm/Group | Intent-to-Treat (ITT) - Secondary Endpoint 4 (R-wave Sensed Amplitude at 6-Mo)
Number analyzed (Participants) | 158
mV | 12.83 (4.78)

11. Secondary Outcome: Pacing Impedance for Solia S Lead at 6 Months
Description: Pacing impedance measurements for Solia S leads implanted in the LBBA at the 6 month follow-up visit.
Time Frame: 6 months post implant
Population: Includes Intent-to-Treat (ITT) subjects with valid pacing impedance measurements at their 6-mo follow-up. Some leads may not have a value at a visit due to valid reasons such as remote due to source documentation being unavailable.
Measure: Mean (Standard Deviation); unit: Impedance (Ω)
Groups:
- Intent-to-Treat (ITT) - Secondary Endpoint 5 (Pacing Impedance at 6-Mo): All enrolled subjects (subjects with successfully implanted Solia S in the LBBA)
Arm/Group | Intent-to-Treat (ITT) - Secondary Endpoint 5 (Pacing Impedance at 6-Mo)
Number analyzed (Participants) | 160
Impedance (Ω) | 526.7 (96.7)

12. Secondary Outcome: Pacing Threshold Measurements for Solia S Lead at 12 Months
Description: Pacing threshold measurements for Solia S leads implanted in the LBBA at the 12 month follow-up visit.
Time Frame: 12 months post implant
Population: Includes Intent-to-Treat (ITT) subjects with valid threshold measurements at their 12-mo follow-up. Some leads may not have a value at a visit due to valid reasons, such as remote threshold information (capture control or automatic threshold measurement) is not available or thresholds not being performed at 0.4 ms, or due to source documentation being unavailable.
Measure: Mean (Standard Deviation); unit: Volts @ 0.4ms
Groups:
- Intent-to-Treat (ITT) - Secondary Endpoint 3 (Pacing Threshold at 12-Mo): All enrolled subjects (subjects with successfully implanted Solia S in the LBBA)
Arm/Group | Intent-to-Treat (ITT) - Secondary Endpoint 3 (Pacing Threshold at 12-Mo)
Number analyzed (Participants) | 144
Volts @ 0.4ms | 0.98 (0.29)

13. Secondary Outcome: Sensing Measurements for Solia S Lead at 12 Months
Description: R-wave sensing amplitude measurements for Solia S leads implanted in the LBBA at the 12 month follow-up visit.
Time Frame: 12 months post implant
Population: Includes Intent-to-Treat (ITT) subjects with valid R-wave sensed amplitude measurements at their 12-mo follow-up. Some leads may not have a value at a visit due to valid reasons, such as atrial fibrillation or complete heart block, or due to source documentation being unavailable.
Measure: Mean (Standard Deviation); unit: mV
Groups:
- Intent-to-Treat (ITT) - Secondary Endpoint 4 (R-wave Sensed Amplitude at 12-Mo): All enrolled subjects (subjects with successfully implanted Solia S in the LBBA)
Arm/Group | Intent-to-Treat (ITT) - Secondary Endpoint 4 (R-wave Sensed Amplitude at 12-Mo)
Number analyzed (Participants) | 152
mV | 12.76 (4.83)

14. Secondary Outcome: Pacing Impedance for Solia S Lead at 12 Months
Description: Pacing impedance measurements for Solia S leads implanted in the LBBA at the 12 month follow-up visit.
Time Frame: 12 months post implant
Population: Includes Intent-to-Treat (ITT) subjects with valid pacing impedance measurements at their 12-mo follow-up. Some leads may not have a value at a visit due to valid reasons such as remote due to source documentation being unavailable.
Measure: Mean (Standard Deviation); unit: Impedance (Ω)
Groups:
- Intent-to-Treat (ITT) - Secondary Endpoint 5 (Pacing Impedance at 12-Mo): All enrolled subjects (subjects with successfully implanted Solia S in the LBBA)
Arm/Group | Intent-to-Treat (ITT) - Secondary Endpoint 5 (Pacing Impedance at 12-Mo)
Number analyzed (Participants) | 155
Impedance (Ω) | 521.8 (96.6)

ADVERSE EVENTS:
Time Frame: Overall study duration of 12 months: from implant (or implant attempt) through each subject's exit date
Description: Adverse events with onset after consent through the study exit date are collected via site review of subject's medical records and subject interview for 1) enrolled subjects and 2) subjects with an unsuccessful implant attempt or implant not meeting success criteria. If a subject is exited as a screen failure after having started the implant procedure, adverse events potentially related to the device or procedure will be collected.
Groups:
- Subjects With a Successful Solia S Implant or Unsuccessful Implant Attempt in the LBBA: This group includes all enrolled subjects (subjects with successfully implanted Solia S in the LBBA) and subjects with an unsuccessful implant attempt of the Solia S in the LBBA.
Arm/Group | Subjects With a Successful Solia S Implant or Unsuccessful Implant Attempt in the LBBA
All-Cause Mortality (participants affected / at risk) | 9/186
Serious Adverse Events (participants affected / at risk) | 52/186
Other Adverse Events (participants affected / at risk) | 0/186
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Subjects With a Successful Solia S Implant or Unsuccessful Implant Attempt in the LBBA (N=186)
Solia S LBBA Lead Related - Lead Dislodgement (Product Issues) | 3 (3)
Procedure Related - Other Implant Procedure Related Adverse Event (Surgical and medical procedures) | 1 (1)
Procedure Related - Deep Vein Thrombosis (Vascular disorders) | 1 (1)
Procedure Related - Infection (Infections and infestations) | 1 (1)
Procedure Related - Hospital Admission for any Reason Attributable to Implant Procedure (Surgical and medical procedures) | 1 (1)
Procedure Related - Pneumo or Hemothorax Associated with Implant Procedure (Injury, poisoning and procedural complications) | 1 (1)
Other Implanted System Related - RA Lead Dislodgement (Product Issues) | 4 (4)
Other Implanted System Related - Other Unexpected Complication Related to RA Lead (Product Issues) | 1 (1)
Other Implanted System Related - Other Pulse Generator Related Adverse Event (Product Issues) | 1 (1)
Other Implanted System Related - Abnormal RA Lead Performance (Product Issues) | 1 (1)
Not Implanted System or Procedure Related - Cardiac Disorders (Cardiac disorders) | 17 (25)
Not Implanted System or Procedure Related - Respiratory, Thoracic, and Mediastinal Disorders (Respiratory, thoracic and mediastinal disorders) | 11 (17)
Not Implanted System or Procedure Related - Surgical and Medical Procedures (Surgical and medical procedures) | 10 (10)
Not Implanted System or Procedure Related - Infections and Infestations (Infections and infestations) | 8 (9)
Not Implanted System or Procedure Related - General Disorders (General disorders) | 8 (8)
Not Implanted System or Procedure Related - Renal and Urinary Disorders (Renal and urinary disorders) | 5 (5)
Not Implanted System or Procedure Related - Gastrointestinal Disorders (Gastrointestinal disorders) | 3 (4)
Not Implanted System or Procedure Related - Hepatobiliary Disorders (Hepatobiliary disorders) | 2 (4)
Not Implanted System or Procedure Related - Vascular Disorders (Vascular disorders) | 4 (4)
Not Implanted System or Procedure Related - Neoplasms Benign, Malignant, and Unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3)
Not Implanted System or Procedure Related - Nervous System Disorders (Nervous system disorders) | 2 (3)
Not Implanted System or Procedure Related - Injury, Poisoning and Procedural Complications (Injury, poisoning and procedural complications) | 2 (2)
Not Implanted System or Procedure Related - Blood and Lymphatic System Disorders (Blood and lymphatic system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After publication of trial results, PIs have the right to publish and/or present the results of the study generated or collected at the institution. The sponsor requires 30 days to review the publication and has the right to obtain input from other investigators in the study. Additionally, the sponsor has the right to delete any confidential information or other proprietary information and may extend the review period if this type of information is included.

DOCUMENTS (3):
  • Study Protocol: Protocol Pages 1-48 (2022-08-10): https://cdn.clinicaltrials.gov/large-docs/63/NCT05251363/Prot_000.pdf
  • Study Protocol: Protocol Pages 49-81 (2022-08-10): https://cdn.clinicaltrials.gov/large-docs/63/NCT05251363/Prot_001.pdf
  • Statistical Analysis Plan (2024-01-19): https://cdn.clinicaltrials.gov/large-docs/63/NCT05251363/SAP_002.pdf